CLINICAL TRIAL: NCT03943186
Title: Non-interventional Study to Investigate the Application of Ectoin Containing Lozenges (EHT02) in Patients With Acute, Viral Pharyngitis.
Brief Title: Application of Ectoin Containing Lozenges (EHT02) in Patients With Acute, Viral Pharyngitis.
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: btph-014-2018-EHT02
Record Dates: First submitted 2019-01-21; First posted 2019-05-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Acute Viral Pharyngitis
Keywords: non-interventional study; Ectoin; Lozenges; Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ectoin Lozenges Honey Lemon: application of 1 Lozenge every three hours or as often as required, not more than 10 lozenges per day
  Interventions: Device: Ectoin Lozenges Honey Lemon
- Hyaluronic acid/Icelandic moss Lozenges: application as often as required, not more than 6 lozenges per day
  Interventions: Device: Hyaluronic Acid/Icelandic moss Lozenges

INTERVENTIONS:
Device: Ectoin Lozenges Honey Lemon — application of Ectoin Lozenges (EHT02) in accordance with the instructions for use
  Other Names: EHT02
  Groups: Ectoin Lozenges Honey Lemon
Device: Hyaluronic Acid/Icelandic moss Lozenges — application of the lozenges in accordance with the instructions for use
  Groups: Hyaluronic acid/Icelandic moss Lozenges

SUMMARY:
The goal of this non-interventional study is to investigate the safety, efficacy and tolerability of Ectoin Lozenges Honey Lemon (EHT02) compared to lozenges containing hyaluronic acid and islandic moss in the treatment of acute viral pharyngitis.

DETAILED DESCRIPTION:
The current non-interventional study aims to investigate the efficacy and tolerability of Ectoin Lozenges Honey Lemon in patients suffering from acute viral pharyngitis. Participants receive treatments as part of routine medical care, and participants can choose one of two treatment options: a) Ectoin Lozenges Honey Lemon or b) lozenges containing hyaluronic acid and icelandic moss.

Efficacy will be studied by documentation of the following symptoms:

* pain on swallowing
* hoarseness
* urge to cough
* dry mouth and throat
* redness of oropharynx and larynx
* sore throat
* impairment of free breathing
* general feeling of illness

In parallel, participating patients will document their symptoms over the entire study duration in patient diaries.

The observation takes place over a period of seven days.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute viral pharyngitis

Exclusion Criteria:

* patients with known intolerance to one of the substances used
* Pregnancy
* Surgical Procedures in the mouth and throat region prior to the study
* Bacterial Pharyngitis
* symptoms in the throat since more than 5 days
* Contraindications according to the instructions for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with acute viral pharyngitis
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-13 (Actual)

PRIMARY OUTCOMES:
Change in Pharyngitis symptom score evaluated by the physician | day 1 and day 7
  The intensity of the symptoms will be graded on a continuous numeric scale, i.e. absent-0, severe-10.
  The following signs and symptoms will be documented:
  * pain on swallowing
  * hoarseness
  * urge to cough
  * dry mouth and throat
  * reddening of oropharynx
  * reddening of larynx
  * sore throat
  * impairment of free breathing
  * patient's general condition

SECONDARY OUTCOMES:
Change in Pharyngitis Symptoms evaluated in patient's diaries | 7 days
  The intensity of the symptoms and signs will be graded on a continuous numeric scale, i.e. absent-0, severe-10.
  The following signs and symptoms will be documented:
  * pain on swallowing
  * hoarseness
  * urge to cough
  * dry mouth and throat
  * sore throat
  * impairment of free breathing
  * patient's general condition
Change of Saliva production evaluated by the physician | day 7
  Assessment on a continuous numeric scale (0-no, 10-yes)
Evaluation how efficient the treatment is judged by physician | day 7
  Assessment on a continuous numeric scale (0-bad, 10-very good)
Evaluation how efficient the treatment is judged by patient | 7 days
  Assessment on a continuous numeric scale (0-bad, 10-very good)
Evaluation how treatment is tolerated (judged by physician) | day 7
  Assessment on a continuous numeric scale (0-bad, 10-very good)
Evaluation how treatment is tolerated (judged by patients) | 7 days
  Assessment on a continuous numeric scale (0-bad, 10-very good)
Evaluation of compliance evaluated by physician | day 7
  Assessment on a continuous numeric scale (0-bad, 10-very good)
Incidence of adverse events/serious adverse events | 7 days
  All occuring adverse events/serious adverse events will be documented during the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Bilstein, Dr, Study Director — CSO
Locations (1):
- bitop AG, Dortmund, Germany

IPD SHARING:
Plan to Share IPD: No